CLINICAL TRIAL: NCT05438095
Title: Medication Adherence and Clinical Outcomes in Sarcoidosis
Brief Title: Medication Adherence in Patients With Sarcoidosis
Acronym: MAPS
Status: Active, not recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00299921; 1K23HL148527-01A1 (NIH)
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Medication Adherence; Sarcoidosis
Keywords: Sarcoidosis; Adherence
MeSH Terms: conditions — Medication Adherence; Sarcoidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collecting blood: Complete Blood Count (CBC) with differential. Will also be collecting Peripheral Blood Mononuclear Cells (PBMCs) and some genetic material will be obtained through these PBMCs.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of the study is to look at the relationship between how individuals with Sarcoidosis take the sarcoidosis medicines and how it affects the disease, to evaluate any factors that may make individuals not want to take the medicines, and to develop and refine ways to help support individuals with Sarcoidosis especially when it comes to the medicines. The overall hypothesis is higher medication adherence will be associated with better clinical outcomes in sarcoidosis. The investigators will enroll 150 patients with biopsy proven pulmonary sarcoidosis for at least one year who are on any oral treatment regimen for at least six months into a 12-month longitudinal study.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Physician diagnosis of Sarcoidosis.
* Biopsy proven pulmonary involvement of Sarcoidosis.
* On oral Sarcoidosis medications for at least 6 months.
* Permanently reside in Maryland or D.C.
* Fully vaccinated against COVID-19.

Exclusion Criteria:

* Non-english speaking.
* Unable to provide consent.
* Unable to participate in orally administered questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals with Sarcoidosis who are seen at the Johns Hopkins Sarcoidosis clinic.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in King's Sarcoidosis Health Questionnaire (KSQ) score | Baseline, 6 months and 12 months
  The KSQ is a 29-item validated measure of sarcoidosis health status. Scores range from 0 to 100. Higher KSQ scores are better. Lower KSQ scores are worse.
Change in St. George's Respiratory Questionnaire (SGRQ) score | Baseline, 6 months and 12 months
  The SGRQ is an instrument that contains 50 items in three subscales (symptoms, activity, and impact). Scores range from 100 to 0. Lower scores for the SGRQ are better and higher scores are worse.
Change in Forced Expiratory Volume (FEV1) as assessed by Pulmonary Function Testing | Baseline, 6 months and 12 months
  Forced Expiratory Volume (FEV1) will be collected by performing Pulmonary Function Testing using spirometry. FEV1 is the maximum amount of air that can be forcibly exhaled in one second.
Change in Forced Vital Capacity (FVC) as assessed by Pulmonary Function Testing | Baseline, 6 months and 12 months
  Forced Vital Capacity (FVC) will be collected by performing Pulmonary Function Testing using spirometry. FVC is the amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible.
Change in Diffusing Capacity of Lung for Carbon Monoxide (DLCO) as assessed by Pulmonary Function Testing | Baseline, 6 months and 12 months
  Diffusing Capacity of Lung for Carbon Monoxide (DLCO) is a measure of the efficiency of lung gas transfer. DLCO will be collected by performing Pulmonary Function Testing after performing spirometry.
Change in 6-minute walk distance | Baseline, 6 months and 12 months
  The distance (in meters) a participant is able to walk in 6 minutes will be assessed.
Change in Modified Medical Research Council Dyspnea Scale (MRC) score | Baseline, 6 months and 12 months
  MRC is a simple scale that has been validated as a method of categorizing patients in terms of their disability attributable to dyspnea. The scale has 5 items on it. Scores range from 0 to 4. Higher scores are worse and lower scores are better.
Change in Health Care Utilization (HCU) as assessed by the CRISP Database | 12 months prior to enrollment and the duration of the study for a total of 24 months
  Health Care Utilization (HCU) for 12 months prior to enrollment and the duration of the study for a total of 24 months will be obtained through the Chesapeake Regional Information System for our Patients (CRISP) database. With consent, researchers are able to receive real-time notifications whenever a participant receives care at any of the hospitals or long-term care facilities. Data available on participants includes records from hospitalizations such as discharge summaries, diagnosis, imaging, and laboratory values. Hospitalization and emergency department (ED) utilization will be coded as a yes/no event. We will also collect self-report hospitalizations and ED visits from the participants at each study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Sharp, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Asthma and Allergy Center, Baltimore, Maryland
  - Johns Hopkins Greenspring Station, Timonium, Maryland